CLINICAL TRIAL: NCT00381901
Title: Protocol of Herceptin Adjuvant With Reduced Exposure, a Randomised Comparison of 6 Months vs 12 Months in All Women Receiving Adjuvant Herceptin [PHARE]
Brief Title: Trastuzumab for 6 Months or 1 Year in Treating Women With Nonmetastatic Breast Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, France (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000509793; INCA-PHARE; INCA-RECF0146; EUDRACT-2006-000070-67
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IA breast cancer; stage IB breast cancer; recurrent breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Amplified Fragment Length Polymorphism Analysis; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: trastuzumab
Genetic: polymorphism analysis
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving trastuzumab for 6 months is as effective as giving trastuzumab for 1 year in treating patients with breast cancer.

PURPOSE: This randomized phase III trial is studying trastuzumab to see how well it works when given for 6 months compared to 12 months in treating women with nonmetastatic breast cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival of women with nonmetastatic, resectable breast cancer treated with adjuvant trastuzumab (Herceptin®) for 6 months vs 12 months.

Secondary

* Compare cardiotoxicity in patients receiving these regimens.
* Compare the cardiotoxicity and disease-free survival of patients receiving concurrent trastuzumab and chemotherapy vs sequential administration.
* Correlate HER-2 polymorphism with disease-free survival/cardiotoxicity in these patients.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center, modality of adjuvant chemotherapy (concurrent vs sequential), and adjuvant hormonal therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control arm, 12-month therapy): Patients continue to receive trastuzumab (Herceptin®) IV until a total of 12 months of therapy is completed in the absence of disease progression or unacceptable toxicity.
* Arm II (experimental arm, 6-month therapy): Patients continue to receive trastuzumab* IV until a total of 6 months of therapy is completed in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who have already finished 6 months of trastuzumab at randomization do not receive further trastuzumab.

Some patients undergo blood collection for HER-2 polymorphism analysis.

After completion of study therapy, patients are followed periodically for approximately 5 years.

PROJECTED ACCRUAL: A total of 7,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast
* Nonmetastatic disease

  * Positive or negative axillary nodes
  * Tumor size ≥ 10 mm
* Resectable disease
* Must have received ≥ 4 courses of chemotherapy for this disease
* A 12-month adjuvant treatment with trastuzumab (Herceptin®) has been initiated

  * Informed consent form must be signed between the third and sixth months of trastuzumab therapy
* Overexpression of HER-2 in the invasive component of the primary tumor as indicated by 1 of the following:

  * 3+ by immunohistochemistry (IHC)
  * 2+ by IHC and confirmation by fluorescent in situ hybridization (FISH) or chromogenic in situ hybridization (CISH)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* LVEF considered favorable for continuing trastuzumab treatment as measured by echocardiography or MUGA at 2-4 months after beginning adjuvant trastuzumab
* No serious cardiac illness or medical condition precluding trastuzumab treatment, including any of the following:

  * History of documented congestive heart failure
  * High-risk uncontrolled arrhythmias
  * Angina pectoris requiring antianginal medication
  * Severe dyspnea at rest or oxygen-dependent
* No known hypersensitivity to trastuzumab, murine proteins, or any of the excipients
* Not pregnant or nursing
* No social, geographical, or psychological condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Other prior anti-HER-2 therapy allowed
* No prior trastuzumab other than initiation of trastuzumab adjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time to recurrence

SECONDARY OUTCOMES:
Cardiotoxicity as measured by LVEF
Distant metastasis-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Pivot, MD, PhD, Study Chair — Hopital Jean Minjoz
Locations (82):
- France (82):
  - Centre Paul Papin, Angers
  - Centre Hospitalier d'Annecy, Annecy
  - Centre Hospitalier La Fontonne, Antibes
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - Institut Sainte Catherine, Avignon
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - C.H.U. de Brest, Brest
  - Centre Hospitalier General, Brivé
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Clinique Notre Dame du Bon Secours, Chartres
  - Hopital Louis Pasteur, Chartres
  - Hopital Antoine Beclere, Clamart
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier de Dax, Dax
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Hopital Jean Monnet, Épinal
  - Hopital Clarac, Fort de France Cedex
  - Institut Prive de Cancerologie, Grenoble
  - Clinique Sainte-Marguerite, Hyères
  - Centre De Radiotherapie Charlebourg, La Garenne-Colombes
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hopital Andre Mignot, Le Chesnay
  - Clinique Victor Hugo, Le Mans
  - Institut d'Oncologie Hartmann, Levallois-Perret
  - Hopital Robert Boulin, Libourne
  - Clinique Chenieux, Limoges
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Medical Parot, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Clinique Claude Bernard, Metz
  - Centre de Radiologie et de Traitement des Tumeurs, Meudon-la-Forêt
  - CH Meulan, Meulan-en-Yvelines
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Montelimar, Montélimar
  - Centre Hospitalier de Montlucon, Montluçon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Clinique Clementville, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Centre Catherine de Sienne, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint-Herblain
  - Clinique Les Genets, Narbonne
  - Clinique Hartmann, Neuilly-sur-Seine
  - Clinique Belvedere, Nice
  - Clinique Saint George, Nice
  - Centre Antoine Lacassagne, Nice
  - C.H.U. de Nimes - Groupe Hospitals-Universitaire Caremeau, Nîmes
  - Clinique De Valdegour, Nîmes
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Curie Hopital, Paris
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Centre Hospitalier - Pau, Pau
  - Clinique Saint - Pierre, Perpignan
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Intercommunal de Poissy, Poissy
  - Hopital Jean Bernard, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - CHG Roanne, Roanne
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Etienne Dolet, Saint-Nazaire
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Clinique Sainte Clotilde, Sainte Clotilde
  - Clinique de l'Orangerie, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Intercommunal Toulon - La Seyne Sur Mer, Toulon
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours

REFERENCES:
- [Derived] Pivot X, Romieu G, Debled M, Pierga JY, Kerbrat P, Bachelot T, Lortholary A, Espie M, Fumoleau P, Serin D, Jacquin JP, Jouannaud C, Rios M, Abadie-Lacourtoisie S, Venat-Bouvet L, Cany L, Catala S, Khayat D, Gambotti L, Pauporte I, Faure-Mercier C, Paget-Bailly S, Henriques J, Grouin JM; PHARE trial investigators. 6 months versus 12 months of adjuvant trastuzumab in early breast cancer (PHARE): final analysis of a multicentre, open-label, phase 3 randomised trial. Lancet. 2019 Jun 29;393(10191):2591-2598. doi: 10.1016/S0140-6736(19)30653-1. Epub 2019 Jun 6. PMID 31178155
- [Derived] Jacquinot Q, Paget-Bailly S, Fumoleau P, Romieu G, Pierga JY, Espie M, Lortholary A, Nabholtz JM, Mercier CF, Pauporte I, Henriques J, Pivot X. Fluctuation of the left ventricular ejection fraction in patients with HER2-positive early breast cancer treated by 12 months of adjuvant trastuzumab. Breast. 2018 Oct;41:1-7. doi: 10.1016/j.breast.2018.06.001. Epub 2018 Jun 15. PMID 29913374
- [Derived] Curtit E, Pivot X, Henriques J, Paget-Bailly S, Fumoleau P, Rios M, Bonnefoi H, Bachelot T, Soulie P, Jouannaud C, Bourgeois H, Petit T, Tennevet I, Assouline D, Mathieu MC, Jacquin JP, Lavau-Denes S, Darut-Jouve A, Ferrero JM, Tarpin C, Levy C, Delecroix V, Trillet-Lenoir V, Cojocarasu O, Meunier J, Pierga JY, Kerbrat P, Faure-Mercier C, Blanche H, Sahbatou M, Boland A, Bacq D, Besse C, Thomas G, Deleuze JF, Pauporte I, Romieu G, Cox DG. Assessment of the prognostic role of a 94-single nucleotide polymorphisms risk score in early breast cancer in the SIGNAL/PHARE prospective cohort: no correlation with clinico-pathological characteristics and outcomes. Breast Cancer Res. 2017 Aug 22;19(1):98. doi: 10.1186/s13058-017-0888-4. PMID 28830573
- [Derived] Pivot X, Fumoleau P, Pierga JY, Delaloge S, Bonnefoi H, Bachelot T, Jouannaud C, Bourgeois H, Rios M, Soulie P, Jacquin JP, Lavau-Denes S, Kerbrat P, Cox D, Faure-Mercier C, Pauporte I, Gligorov J, Curtit E, Henriques J, Paget-Bailly S, Romieu G. Superimposable outcomes for sequential and concomitant administration of adjuvant trastuzumab in HER2-positive breast cancer: Results from the SIGNAL/PHARE prospective cohort. Eur J Cancer. 2017 Aug;81:151-160. doi: 10.1016/j.ejca.2017.05.020. Epub 2017 Jun 16. PMID 28624696
- [Derived] Pivot X, Suter T, Nabholtz JM, Pierga JY, Espie M, Lortholary A, Khayat D, Pauporte I, Romieu G, Kramar A, Fumoleau P. Cardiac toxicity events in the PHARE trial, an adjuvant trastuzumab randomised phase III study. Eur J Cancer. 2015 Sep;51(13):1660-6. doi: 10.1016/j.ejca.2015.05.028. Epub 2015 Jul 7. PMID 26163096
- [Derived] Kramar A, Bachelot T, Madrange N, Pierga JY, Kerbrat P, Espie M, Fumoleau P, Pauporte I, Khayat D, Romieu G, Pivot X. Trastuzumab duration effects within patient prognostic subgroups in the PHARE trial. Ann Oncol. 2014 Aug;25(8):1563-70. doi: 10.1093/annonc/mdu177. Epub 2014 May 14. PMID 24827132
- [Derived] Pivot X, Romieu G, Debled M, Pierga JY, Kerbrat P, Bachelot T, Lortholary A, Espie M, Fumoleau P, Serin D, Jacquin JP, Jouannaud C, Rios M, Abadie-Lacourtoisie S, Tubiana-Mathieu N, Cany L, Catala S, Khayat D, Pauporte I, Kramar A; PHARE trial investigators. 6 months versus 12 months of adjuvant trastuzumab for patients with HER2-positive early breast cancer (PHARE): a randomised phase 3 trial. Lancet Oncol. 2013 Jul;14(8):741-8. doi: 10.1016/S1470-2045(13)70225-0. Epub 2013 Jun 11. PMID 23764181